CLINICAL TRIAL: NCT00485784
Title: Interest of Circulating Endothelial Biomarkers in Vascular Pregnancy Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006/26
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Pre-Eclampsia
Keywords: Identify in a population of patients with a PE, an IUGR and a FD a modification of circulating endothelial biomarkers compared with normal pregnancy.
MeSH Terms: conditions — Pre-Eclampsia | interventions — Hematologic Tests

ARMS (4):
- control group (Sham Comparator): control group
  Interventions: Other: Blood test
- prééclampsies group (Experimental): prééclampsies group
  Interventions: Other: Blood test
- RCIU group (Experimental): RCIU group
  Interventions: Other: Blood test
- MFIU group (Experimental): MFIU group
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Blood test

SUMMARY:
This is a prospective multicentric study including four clinical units of Gynecology and Obstetrics (3 public health hospitals and one private team), one research team in Hematology and one Center of Clinical investigation (CIC).

The objective is to identify, beside the pregnancy, in a population of patients with a preeclampsia (PE), with fetus presenting with growth restriction (IUGR) and a fetal demise (FD) a modification of circulating endothelial biomarkers compared with normal pregnancy.

We want to understand better the physiopathology of preeclampsia and propose to patients with an endothelial dysfunction a early prevention of preeclampsia.

Patients will be tested 3 times : At the pregnancy events; then 8 weeks and 12 months after the birth.

Four groups will be constituted among patients: PE, IUGR, FD and normal pregnancy.

Normal pregnancy will be tested as controls. The next pregnancy presenting in the unit to medical pregnancy follow up will be invited to participate.

The main judgment criteria will be the levels of endothelial microparticles 8 weeks after the event.

The study will last 3 years. The number of patient to include is 280.

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients aged more than 18 years and more than 12 weeks of gestation for FD group, 20 weeks of gestation for PE or IUGR group , presenting either:
* PE (arterial pressure more than 140 mm Hg and 90 mm Hg) and at least a proteinuria evaluated on stick (one point) or 300 mg/24h.
* IUGR with biometries below 5° percentile according to the graphs of fetal echography college after 20 weeks of gestation.
* FD after 12 weeks of gestation or with a cranio-caudal length of more than 45 mm.
* Normal pregnancy adjusted for gestational age and parity : Patient should have no cardio-vascular past with a normal complication at the inclusion time and from which pregnancy remains uneventful until the term. The onset of premature delivery, hypertension or fetal growth restriction will exclude patients from the control group.
* social security cover
* written informed consent

Exclusion Criteria:

* Foetal malformation
* APLS known
* Set back of patient consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2007-07; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Bring to light except the pregnancy within a population of presenting patients one EP, a RCIU and a MFIU a modification of biomarkers circulating endothéliaux with regard to the normal pregnancy. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRETELLE, PU-PH, Principal Investigator — Unité Mère-Enfant Hôpital Nord 13005 Marseille - Assistance Publique Hôpitaux de Marseille
Locations (4):
- France (4):
  - Hôpital Saint-Joseph - Service de Gynécologie-Obstétrique, Marseille
  - Hôpital Nord, Marseille
  - Hôpital de la Conception, Marseille
  - Chu Nice Hopital de L'Archet, Nice